CLINICAL TRIAL: NCT03633695
Title: Clinical Evaluation of a Small Aperture Extended Depth of Focus Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAIL-101-UNI
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: Cataract; Presbyopia
Keywords: Cataract; Intraocular lens
MeSH Terms: conditions — Cataract; Presbyopia | interventions — Lenses, Intraocular; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Examiner masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- IC-8 IOL Group (Experimental): A monofocal IOL (TECNIS ZCB00, ZCT150 or ZCT225 or AcrySof IQ SA60WF, SA6AT3 or SA6AT4) implanted in the first eye. The AcuFocus IC-8 IOL implanted in the second eye.
  Interventions: Device: IC-8 IOL Group
- Control Group (Active Comparator): A monofocal IOL (TECNIS ZCB00, ZCT150 or ZCT225 or AcrySof IQ SA60WF, SA6AT3 or SA6AT4) bilaterally implanted.
  Interventions: Device: Control Group

INTERVENTIONS:
Device: IC-8 IOL Group — A monofocal IOL (TECNIS ZCB00, ZCT150 or ZCT225 or AcrySof IQ SA60WF, SA6AT3 or SA6AT4) implanted in the first eye for use over the lifetime of the patient. The IC-8 IOL implanted in the second eye for use over the lifetime of the patient.
  Other Names: Intraocular Lens
  Arms: IC-8 IOL Group
Device: Control Group — A monofocal IOL (TECNIS ZCB00, ZCT150 or ZCT225 or AcrySof IQ SA60WF, SA6AT3 or SA6AT4) bilaterally implanted for lifetime use of the patient.
  Other Names: Intraocular lens
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the IC-8 IOL implanted in one eye and a monofocal or monofocal toric IOL implanted in the fellow eye in accordance with the indication.

DETAILED DESCRIPTION:
Eligible patients will complete up to 12 study visits over a 12-month period. All subjects will complete a preoperative examination of both eyes to assess study eligibility: operative visit (each eye) and up to 9 postoperative visits (Day 1 - each eye, Week 1 - each eye, Month 1 - each eye or combined, Month 3 - both eyes, Month 6 - both eyes, and Month 12 - both eyes). The first eye must meet specific qualification criteria in order to proceed with IOL implantation in the second eye. The second eye should be implanted within 45 days of the first eye.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 22 years of age;
2. Able to comprehend and have signed a statement of informed consent;
3. Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits;
4. Planned crystalline lens removal by phacoemulsification, with or without femtosecond laser-assisted extraction, and posterior chamber IOL implantation in both eyes;
5. Cataractous lens changes as demonstrated by best-corrected visual acuity (BCDVA) of 20/40 or worse either with or without a glare source present;
6. Potential for postoperative BCDVA of 20/25 or better in each eye
7. Clear intraocular media, other than cataract.

Exclusion Criteria:

1. Requiring an IC-8 intraocular lens outside the available spherical power range
2. Pharmacologically dilated pupil size less than 6 mm in either eye;
3. Inability to achieve stable keratometric readings for contact lens wearers
4. Irregular astigmatism in either eye;
5. Preoperative corneal astigmatism > 1.50 diopters in either eye
6. Active or recurrent anterior segment pathology
7. Presence of ocular abnormalities other than cataract as specified in the protocol
8. Diagnosis of dry eye in which patients are unable to maintain eye comfort or adequate vision even with dry eye medication;
9. Congenital cataracts;
10. Previous corneal or intraocular surgery
11. History of ocular trauma or ocular conditions expected to require retinal laser treatment or other surgical intervention;
12. Systemic conditions as specified in the protocol;
13. Patient is pregnant, plans to become pregnant, or is lactating
14. Concurrent participation or participation in any clinical trial up to 30 days prior to preoperative visit.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magda Michna, PhD, Study Director — AcuFocus, Inc.
Locations (21):
- United States (21):
  - Fishkind, Bakewell, Maltzman, Hunter & Associates Eye Care & Surgery Center, Tucson, Arizona
  - Empire Eye & Laser Center, Bakersfield, California
  - Harvard Eye Associates, Laguna Hills, California
  - Altos Eye Physicians, Los Altos, California
  - Advanced Vision Care, Los Angeles, California
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Eye Center of North Florida, Panama City, Florida
  - Chu Vision Institute, Bloomington, Minnesota
  - Pepose Vision Institute, St Louis, Missouri
  - Kugler Vision, Omaha, Nebraska
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Physicians Protocol, Greensboro, North Carolina
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Bucci Laser Vision, Wilkes-Barre, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Hoopes Vision, Draper, Utah
  - Utah Eye Centers, Ogden, Utah
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vukich J, Thompson V, Yeu E, Wiley WF, Bafna S, Koch DD, Lin L, Michna M. Evaluating the small aperture intraocular lens: depth of focus and the role of refraction and preoperative corneal astigmatism in visual performance. J Cataract Refract Surg. 2024 Nov 1;50(11):1165-1172. doi: 10.1097/j.jcrs.0000000000001524. PMID 39075732
- See also: Sponsor website — http://www.acufocus.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 21 investigative sites within the United States from 04 December 2018 to 21 August 2019. The investigative sites were comprised of similar clinic, surgical center, and equipment requirements necessary for the intended use of the IC-8™ IOL.
Pre-assignment Details: A total of 548 subjects signed the informed consent form, 79 of whom did not meet inclusion/exclusion criteria and were considered screen failures; leaving 469 subjects who were considered provisionally enrolled in the study. A total of 16 subjects were disqualified or discontinued from the study prior to second eye implantation. There were 453 subjects who were successfully bilaterally implanted in the study (reporting group).
Units Other Than Participants: Eyes
Groups:
- IC-8™ IOL Group: Subjects implanted with a monofocal IOL (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the first eye and the IC-8™ Intraocular Lens (IOL) in the second eye.
  * Subjects in this Group were assigned to Astigmatism Group 1 (<1.0 D) or Astigmatism Group 2 (1.0 D - 1.5 D), as determined by preoperative corneal astigmatism in the 2nd eye (study eye).
- Control Group: Subjects bilaterally implanted with monofocal IOLs (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOLs (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225).
  * Subjects in this Group were assigned to Astigmatism Group 1 (<1.0 D) or Astigmatism Group 2 (1.0 D - 1.5 D), as determined by preoperative corneal astigmatism in the 2nd eye (fellow eye).
Period: Overall Study
Arm/Group | IC-8™ IOL Group | Control Group
Started | 343; 686 Eyes | 110; 220 Eyes
Astigmatism Group 1 (IC-8™ IOL Group) | 273; 546 Eyes | 0; 0 Eyes
Astigmatism Group 2 (IC-8™ IOL Group) | 70; 140 Eyes | 0; 0 Eyes
Astigmatism Group 1 (Control Group) | 0; 0 Eyes | 91; 182 Eyes
Astigmatism Group 2 (Control Group) | 0; 0 Eyes | 19; 38 Eyes
Completed | 331; 662 Eyes | 101; 202 Eyes
Not Completed | 12; 24 Eyes | 9; 18 Eyes
Not completed — Lost to Follow-up | 4 | 5
Not completed — Discontinued | 8 | 4

BASELINE CHARACTERISTICS:
Population: The analysis population includes all eyes with successful bilateral implantation (Intent-to-Treat analysis population). Baseline characteristics were analyzed by subject.
Groups:
- IC-8™ IOL Group: Subjects implanted with a monofocal IOL (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the first eye and the IC-8™ Intraocular Lens (IOL) in the second eye.
- Control Group: Subjects bilaterally implanted with monofocal IOLs (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOLs (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225).
- Total: Total of all reporting groups
Arm/Group | IC-8™ IOL Group | Control Group | Total
Number analyzed (Participants) | 343 | 110 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (7.96) | 69.1 (8.63) | 66.8 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 76 | 287
  Male | 132 | 34 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 10 | 32
  Not Hispanic or Latino | 320 | 100 | 420
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Entries of 'Unknown' or 'Not Reported' represent race reported as 'Other'. During the clinical study there were no participants with 'Unknown' or 'Not Reported' race.
  Participants
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 3 | 3 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 22 | 6 | 28
    White | 311 | 99 | 410
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 6 | 1 | 7
Preoperative Corneal Astigmatism [Count of Participants; unit: Participants] — Each study group (IC-8™ IOL Group, Control Group) included two astigmatism groups, Astigmatism Group 1 (<1.0 D) and Astigmatism Group 2 (1.0 D - 1.5 D). The enrollment ratio was approximately 5:1 for Astigmatism Group 1 vs. Astigmatism Group 2. Subject assignment to Astigmatism Group 1 or Astigmatism Group 2 was determined by preoperative corneal astigmatism in the second eye as measured by optical biometry.
  Participants
    Astigmatism Group 1 (<1.0 D) | 273 | 91 | 364
    Astigmatism Group 2 (1.0 D - 1.5 D) | 70 | 19 | 89

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Photopic Uncorrected Intermediate (66 cm) Visual Acuity (UCIVA)
Description: Visual acuity (VA) was tested binocularly (both eyes) at a distance of 66 cm, without manifest refraction, using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart presenting on a self-calibrating monitor in a computerized testing system. Visual acuity was measured in logarithm of the minimum angle of resolution (logMAR), with a 0.02 logMAR increment corresponding to a single letter on the ETDRS chart.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: For this outcome measure, the number of participants/eyes from the Intent-to-Treat (ITT) population (all subjects who were fully enrolled and were binocularly implanted in the study) that were available for analysis at 6 Months was used. It was pre-specified that results were not separated by Astigmatism Groups for this measure.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 335 | 100
Number analyzed (Eyes) | 670 | 200
logMAR | 0.051 (0.1629) | 0.228 (0.1646)
Statistical Analysis 1: Comparison: IC-8™ IOL Group vs Control Group; The null hypothesis was that the mean acuity for the IC-8 Group was greater (i.e. worse) than or equal to that for the Control Group. The alternative hypothesis was that the mean for the IC-8 Group less (i.e., better) than that for the Control Group; Test type: Superiority; p < .0001, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.177, 95% CI 2-sided [-0.214 to -0.140] — Acuity Difference = IC-8 Group - Control Group

2. Primary Outcome: Mean Binocular Photopic Uncorrected Near (40 cm) Visual Acuity (UCNVA)
Description: Visual acuity (VA) was tested binocularly (both eyes) at a distance of 40 cm, without manifest refraction, using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart presenting on a self-calibrating monitor in a computerized testing system. Visual acuity was measured in logarithm of the minimum angle of resolution (logMAR), with a 0.02 logMAR increment corresponding to a single letter on the ETDRS chart.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 335 | 100
Number analyzed (Eyes) | 670 | 200
logMAR | 0.186 (0.1425) | 0.377 (0.1576)
Statistical Analysis 1: Comparison: IC-8™ IOL Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.191, 95% CI 2-sided [-0.223 to -0.158] — Acuity Difference = IC-8 Group - Control Group

3. Primary Outcome: Mean Binocular Photopic Uncorrected Distance (4 m) Visual Acuity (UCDVA)
Description: Visual acuity (VA) was tested binocularly (both eyes) at a distance of 4 m, with +0.25 D infinity adjustment lens in front of the eyes, using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart presenting on a self-calibrating monitor in a computerized testing system. Visual acuity was measured in logarithm of the minimum angle of resolution (logMAR), with a 0.02 logMAR increment corresponding to a single letter on the ETDRS chart.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 335 | 100
Number analyzed (Eyes) | 670 | 200
logMAR | -0.010 (0.1063) | 0.002 (0.0992)
Statistical Analysis 1: Comparison: IC-8™ IOL Group vs Control Group; The null hypothesis was that the mean acuity for the IC-8 IOL Group is inferior to the Control Group by 0.1 logMAR or more. The alternative hypothesis was that the mean acuity for the IC-8 IOL group is inferior to the Control Group by less than 0.1 logMAR; Test type: Non-Inferiority — Non-inferiority margin was 0.1 logMAR; p < .0001, t-test, 1 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.012, 95% CI 1-sided [upper limit 0.007] — Acuity Difference = IC-8 IOL Group - Control Group

4. Primary Outcome: Mean Monocular Photopic Distance-Corrected Intermediate (66 cm) Visual Acuity (DCIVA) in IC-8™ IOL Eyes
Description: Visual acuity (VA) was tested monocularly (each eye) at a distance of 66 cm, with the distance manifest refraction (with infinity adjustment) in place for that eye, using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart presenting on a self-calibrating monitor in a computerized testing system. Visual acuity was measured in logarithm of the minimum angle of resolution (logMAR), with a 0.02 logMAR increment corresponding to a single letter on the ETDRS chart.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- IC-8™ IOL Eyes (IC-8™ IOL Group): Eyes implanted with the IC-8™ Intraocular Lens (IOL).
- Fellow Eyes (IC-8™ IOL Group): Eyes implanted with a monofocal IOL (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225).
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 335 | 335
Number analyzed (Eyes) | 335 | 335
logMAR | 0.144 (0.1709) | 0.325 (0.1687)
Statistical Analysis 1: Comparison: IC-8™ IOL Eyes (IC-8™ IOL Group) vs Fellow Eyes (IC-8™ IOL Group); The null hypothesis was that the mean acuity for the IC-8 IOL eyes is greater (i.e., worse) than or equal to that for the fellow eyes. The alternative hypothesis was that the mean for the IC-8 IOL eyes is less (i.e., better) than that for the fellow eyes; Test type: Superiority; p < .0001, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.180, 95% CI 2-sided [-0.198 to -0.163] — Acuity Difference = IC-8 IOL Eye (IC-8 IOL Group) - Fellow Eye (IC-8 IOL Group)

5. Primary Outcome: Mean Monocular Photopic Depth of Focus (DOF) in IC-8™ IOL Eyes
Description: Depth of focus was performed monocularly in the IC-8™ IOL Group at the far to near range of vision (+2.00 to -5.00 D), using 100% contrast ETDRS charts in a computerized testing system calibrated for a 4 m test distance, with manifest refraction (no infinity adjustment) in place for the eye(s) being tested. The defocus power was progressively introduced in 0.50 D increments from +2.00 D to +0.50 D and from -0.50 D to -5.00 D, then in 0.25 D increments from +0.50 D to -0.50 D, while visual acuity was measured at each successive defocus step. The depth of focus was estimated as the defocus range between zero defocus and the first point on the negative lens induced mean defocus curve that crosses the 0.2 logMAR using a linear interpolation.
Time Frame: 3 Months (60-110 days post second eye operative visit)
Population: For this outcome measure, the number of participants/eyes from the Intent-to-Treat (ITT) population (all subjects who were fully enrolled and were binocularly implanted in the study) that were available for analysis at 3 Months was used. It was pre-specified that results were not separated by Astigmatism Groups for this measure.
Measure: Mean (Standard Deviation); unit: Diopter
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 335 | 335
Number analyzed (Eyes) | 335 | 335
Diopter | -1.99 (NA) — The negative intercept (outcome measure) was calculated from the means of the two defocus steps where the defocus curve crosses the 0.2 logMAR threshold. | -1.08 (NA) — The negative intercept (outcome measure) was calculated from the means of the two defocus steps where the defocus curve crosses the 0.2 logMAR threshold.
Statistical Analysis 1: Comparison: IC-8™ IOL Eyes (IC-8™ IOL Group) vs Fellow Eyes (IC-8™ IOL Group); Test type: Other; Difference in depth of focus = 0.91 — Difference in depth of focus [IC-8™ IOL Eyes (IC-8™ IOL Group) - Fellow Eyes (IC-8™ IOL Group)]

6. Primary Outcome: Mean Monocular Best-corrected Distance (4 m) Visual Acuity (BCDVA)
Description: Visual acuity (VA) was tested monocularly (each eye) at a distance of 4 m, in photopic conditions, with manifest refraction in place (no infinity adjustment) using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart presenting on a self-calibrating monitor in a computerized testing system. Visual acuity was measured in logarithm of the minimum angle of resolution (logMAR), with a 0.02 logMAR increment corresponding to a single letter on the ETDRS chart.
Time Frame: 12 Months (300-420 days post second eye operative visit)
Population: For this outcome measure, the safety analysis set was used, which, included available data from all eyes that were bilaterally implanted, or for whom implantation of an IC-8™ IOL was attempted (the IC-8 IOL touched the eye during surgery). The Safety and ITT populations were identical in this study. Data from participants/eyes available for analysis at 12 Months was used. It was pre-specified that results were not separated by Astigmatism Groups for this outcome measure.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 331 | 331
Number analyzed (Eyes) | 331 | 331
logMAR | 0.009 (0.1131) | -0.059 (0.0928)
Statistical Analysis 1: Comparison: IC-8™ IOL Eyes (IC-8™ IOL Group) vs Fellow Eyes (IC-8™ IOL Group); The null hypothesis was that the mean acuity for the IC-8 IOL eyes was inferior to the fellow eyes by 0.1 logMAR or more. The alternative hypothesis was that the mean acuity for the IC-8 eyes was inferior to the fellow eyes by less than 0.1 logMAR; Test type: Non-Inferiority — The non-inferiority margin was 0.1 logMAR; p < .0001, t-test, 1 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.068, 95% CI 1-sided [upper limit 0.082] — Acuity Difference = IC-8 IOL Eyes (IC-8 Group) - Fellow Eyes (IC-8 Group)

7. Primary Outcome: Proportion of IC-8™ IOL Eyes Achieving Best-corrected Distance Visual Acuity (BCDVA) 0.3 logMAR or Better Compared to the Safety and Performance Endpoints (SPE) Rates
Description: as for outcome 6
Time Frame: 12 Months (300-420 days post second eye operative visit)
Population: as for outcome 6
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 331 | 331
Number analyzed (Eyes) | 331 | 331
Eyes | 326 | 330

8. Primary Outcome: Proportion of Best-Case IC-8™ IOL Eyes Achieving Best-corrected Distance Visual Acuity (BCDVA) 0.3 logMAR or Better Compared to the Safety and Performance Endpoints (SPE) Rates
Description: Visual acuity (VA) was tested monocularly (each eye) at a distance of 4 m, in photopic conditions, with manifest refraction in place (no infinity adjustment) using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart presenting on a self-calibrating monitor in a computerized testing system. Visual acuity was measured in logarithm of the minimum angle of resolution (logMAR), with a 0.02 logMAR increment corresponding to a single letter on the ETDRS chart. Monocular BCDVA for the IC-8™ IOL eyes of subjects in the Best-Case population was compared to the safety and performance endpoints (SPE) rate for posterior chamber IOLs.
Time Frame: 12 Months (300-420 days post second eye operative visit)
Population: For this outcome measure, the Best-Case analysis was used, which, included subjects with no preoperative ocular pathology, no macular degeneration detected at any time, and no previous surgery for the correction of refractive errors (as defined by ISO 11979-1:2012), as well as no significant macular pathology at any time. Data from participants/eyes available for analysis at 12 Months was used. It was pre-specified that results were not separated by Astigmatism Groups for this outcome measure.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 319 | 319
Number analyzed (Eyes) | 319 | 319
Eyes | 315 | 318

9. Primary Outcome: Rates of IC-8™ IOL Eyes With Cumulative Ocular Serious Adverse Events
Description: The rates of cumulative ocular serious adverse events (SAEs) for IC-8™ IOL eyes were calculated from the time of second eye (IC-8™ IOL eye) implantation through Month 12.
Time Frame: Through 12 Months (300-420 days post second eye operative visit)
Population: as for outcome 6
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 343 | 343
Number analyzed (Eyes) | 343 | 343
Eyes
  Cystoid Macular Edema | 5 | 4
  Hypopyon | 0 | 0
  Endophthalmitis | 1 | 0
  Lens Dislocated from Posterior Chamber | 0 | 0
  Pupillary Block | 0 | 0
  Retinal Detachment | 0 | 0
  Modified Paracentesis | 4 | 3
  Intravitreal Injection | 1 | 1
  Laser Retinopexy | 0 | 1
  Other: Retinal Vein Occlusion | 1 | 0
  Vitrectomy | 4 | 1
  Removal of retained cortex | 2 | 0
  IOL repositioning | 1 | 1

10. Primary Outcome: Rates of IC-8™ IOL Eyes With Cumulative Postoperative Ocular Adverse Events (Secondary Surgical Interventions)
Description: The rates of cumulative ocular adverse events for IC-8™ IOL eyes were calculated from the time of second eye (IC-8™ IOL eye) implantation through Month 12.
Time Frame: Through 12 Months (300-420 days post second eye operative visit)
Population: as for outcome 6
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- IC-8 IOL Eyes (IC-8™ IOL Group): Eyes implanted with the IC-8™ Intraocular Lens (IOL).
- Second Eyes (Control Group); First Eyes (Control Group): Eyes implanted with a monofocal IOL (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOLs (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225).
Arm/Group | IC-8 IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group) | Second Eyes (Control Group) | First Eyes (Control Group)
Number analyzed (Participants) | 343 | 343 | 110 | 110
Number analyzed (Eyes) | 343 | 343 | 110 | 110
Eyes
  Intravitreal Injection | 1 | 1 | 0 | 1
  IOL Exchange | 0 | 0 | 1 | 1
  IOL Repositioning | 1 | 1 | 0 | 1
  Iris Reposition | 0 | 0 | 0 | 1
  Laser Retinopexy | 0 | 1 | 0 | 0
  Laser Vitreolysis | 0 | 0 | 1 | 0
  Modified Paracentesis | 4 | 3 | 0 | 1
  Removal of Retained Cortex | 2 | 0 | 0 | 0
  Vitrectomy | 4 | 1 | 0 | 0

11. Primary Outcome: Rates of IC-8™ IOL Eyes With Persistent Ocular Serious Adverse Events
Description: The rates of persistent (defined as being unresolved at final scheduled visit) ocular adverse events (AEs) for IC-8™ IOL eyes were calculated from the time of second eye (IC-8™ IOL eye) implantation through Month 12.
Time Frame: Through 12 Months (300-420 days post second eye operative visit)
Population: as for outcome 6
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 331 | 331
Number analyzed (Eyes) | 331 | 331
Eyes
  Corneal Stromal Edema | 0 | 0
  Cystoid Macular Edema | 1 | 1
  Iritis | 2 | 1
  Raised IOP Requiring Treatment | 0 | 0
  Other: Retinal Vein Occlusion | 1 | 0

12. Primary Outcome: Rates of IC-8™ IOL Eyes With IC-8™ IOL Removals
Description: as for outcome 10
Time Frame: Through 12 Months (300-420 days post second eye operative visit)
Population: as for outcome 6
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Second Eye (Control Group); First Eye (Control Group): Eyes implanted with an AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00, or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the Control Group.
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group) | Second Eye (Control Group) | First Eye (Control Group)
Number analyzed (Participants) | 343 | 343 | 110 | 110
Number analyzed (Eyes) | 343 | 343 | 110 | 110
Eyes | 0 | 0 | 1 | 1

13. Primary Outcome: Rates of Eyes With Postoperative Ocular Adverse Events (Other Than Secondary Surgical Intervention), Related to Device (Serious and Non-Serious Combined)
Description: The rates of cumulative ocular adverse events (AEs) for IC-8™ IOL eyes were calculated from the time of second eye (IC-8™ IOL eye) implantation through Month 12.
Time Frame: Through 12 Months (300-420 days post second eye operative visit)
Population: as for outcome 6
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- IC-8 IOL Eyes (IC-8™ IOL Group: Eyes implanted with the IC-8™ Intraocular Lens (IOL).
- Fellow Eyes (IC-8™ IOL Group: Eyes implanted with a monofocal IOL (AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00), or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225).
Arm/Group | IC-8 IOL Eyes (IC-8™ IOL Group | Fellow Eyes (IC-8™ IOL Group | Second Eyes (Control Group) | First Eyes (Control Group)
Number analyzed (Participants) | 343 | 343 | 110 | 110
Number analyzed (Eyes) | 343 | 343 | 110 | 110
Eyes
  Device Damage | 1 | 0 | 0 | 0
  Posterior Capsule Opacification | 3 | 1 | 0 | 0
  Altered Visual Depth Perception | 1 | 1 | 0 | 0
  Dysphotopsia | 5 | 3 | 0 | 1
  Halo Vision | 2 | 0 | 0 | 0
  Vision Blurred | 2 | 1 | 0 | 0

14. Secondary Outcome: Tolerance to Preoperative Corneal Astigmatism in IC-8™ IOL Eyes With BCDVA 20/25 at 3 Months
Description: Uncorrected-distance visual acuity (UCDVA) in IC-8™ IOL eyes achieving best-corrected distance visual acuity (BCDVA) of 20/25 or better was compared between eyes with preoperative corneal astigmatism < 1.0 D to eyes with 1.0 D to 1.5 D of preoperative corneal astigmatism.
Time Frame: 3 Months (60-110 days post second eye operative visit)
Population: For this outcome measure, the number of participants/eyes from the modified Intent-to-Treat (mITT) population (subjects from the intent to treat population that achieved BCDVA 20/25 or better) that were available for analysis at 3 Months was used. It was pre-specified that results were not separated by Astigmatism Groups for this measure.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- IC-8™ IOL Eyes With Astigmatism <1.0 D (IC-8™ IOL Group): Eyes with <1.0 D preoperative corneal astigmatism implanted with the IC-8™ Intraocular Lens (IOL).
- IC-8™ IOL Eyes With Astigmatism 1.0 D - 1.5 D (IC-8™ IOL Group): Eyes with 1.0 D - 1.5 D preoperative corneal astigmatism implanted with the IC-8™ Intraocular Lens (IOL).
Arm/Group | IC-8™ IOL Eyes With Astigmatism <1.0 D (IC-8™ IOL Group) | IC-8™ IOL Eyes With Astigmatism 1.0 D - 1.5 D (IC-8™ IOL Group)
Number analyzed (Participants) | 244 | 65
Number analyzed (Eyes) | 244 | 65
logMAR | 0.085 (0.1269) | 0.108 (0.1208)
Statistical Analysis 1: Comparison: IC-8™ IOL Eyes With Astigmatism <1.0 D (IC-8™ IOL Group) vs IC-8™ IOL Eyes With Astigmatism 1.0 D - 1.5 D (IC-8™ IOL Group); The null hypothesis was that the mean acuity in Astigmatism Group 2 was inferior to the Astigmatism Group 1 by 0.12 logMAR or more. The alternative hypothesis was that the mean acuity in Astigmatism Group 2 was inferior to Astigmatism Group 1 by less than 0.12 logMAR; Test type: Non-Inferiority — Non-inferiority margin was 0.12 logMAR; p < .0001, t-test, 1 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.023

15. Secondary Outcome: Mean Monocular Photopic Contrast Sensitivity Without Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested monocularly (each eye) in photopic (well-lit) conditions, without a glare source, using sine waving gratings in a computerized testing system. The photopic spatial frequencies tested were 3, 6, 12, 18 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better contrast sensitivity results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: A subgroup of subjects from the IC-8™ IOL Group (262 enrolled) and Control Group (68 enrolled) available for analysis at 6 Months. It was pre-specified that results were not separated by Astigmatism Groups for this outcome measure.
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 260 | 260
Number analyzed (log units) | 260 | 260
log units on a scale
  Spatial Frequency 3 cpd | 1.935 (0.3768) | 2.202 (0.2542)
  Spatial Frequency 6 cpd | 1.795 (0.3736) | 2.055 (0.3576)
  Spatial Frequency 12 cpd | 1.308 (0.4186) | 1.554 (0.4530)
  Spatial Frequency 18 cpd | 0.832 (0.3996) | 1.072 (0.4220)

16. Secondary Outcome: Mean Monocular Photopic Contrast Sensitivity With Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects, and was tested monocularly (each eye) in photopic (well-lit) conditions, with a glare source, using sine waving gratings in a computerized testing system. The photopic spatial frequencies tested were 3, 6, 12, 18 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 260 | 260
log units on a scale
  Spatial Frequency 3 cpd | 1.620 (0.4219) | 1.822 (0.4247)
  Spatial Frequency 6 cpd | 1.513 (0.3926) | 1.747 (0.4136)
  Spatial Frequency 12 cpd | 1.106 (0.4149) | 1.345 (0.4315)
  Spatial Frequency 18 cpd | 0.659 (0.4161) | 0.887 (0.4171)

17. Secondary Outcome: Mean Monocular Mesopic Contrast Sensitivity Without Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested monocularly (each eye) in mesopic (low-light) conditions, without a glare source, using sine waving gratings in a computerized testing system. The mesopic spatial frequencies tested were 1.5, 3, 6, 12 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 260 | 260
Number analyzed (log units) | 260 | 260
log units on a scale
  Spatial Frequency 1.5 cpd | 1.385 (0.3596) | 1.850 (0.3849)
  Spatial Frequency 3 cpd | 1.475 (0.3882) | 1.964 (0.3662)
  Spatial Frequency 6 cpd | 1.217 (0.3901) | 1.609 (0.4300)
  Spatial Frequency 12 cpd | 0.620 (0.3739) | 0.913 (0.4105)

18. Secondary Outcome: Mean Monocular Mesopic Contrast Sensitivity With Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested monocularly (each eye) in mesopic (low-light) conditions, with a glare source, using sine waving gratings in a computerized testing system. The mesopic spatial frequencies tested were 1.5, 3, 6, 12 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Eyes (IC-8™ IOL Group) | Fellow Eyes (IC-8™ IOL Group)
Number analyzed (Participants) | 260 | 260
Number analyzed (log units) | 260 | 260
log units on a scale
  Spatial Frequency 1.5 cpd | 1.044 (0.4063) | 1.338 (0.4212)
  Spatial Frequency 3 cpd | 1.201 (0.4142) | 1.552 (0.4468)
  Spatial Frequency 6 cpd | 1.035 (0.4337) | 1.353 (0.4224)
  Spatial Frequency 12 cpd | 0.496 (0.3886) | 0.749 (0.4305)

19. Secondary Outcome: Mean Binocular Photopic Contrast Sensitivity Without Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested binocularly (both eyes) in photopic (well-lit) conditions, without a glare source, using sine waving gratings in a computerized testing system. The photopic spatial frequencies tested were 3, 6, 12, 18 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 260 | 67
Number analyzed (log units) | 260 | 67
log units on a scale
  Spatial Frequency 3 cpd | 2.233 (0.2536) | 2.287 (0.1896)
  Spatial Frequency 6 cpd | 2.119 (0.3293) | 2.141 (0.3177)
  Spatial Frequency 12 cpd | 1.689 (0.4263) | 1.654 (0.5124)
  Spatial Frequency 18 cpd | 1.164 (0.4123) | 1.090 (0.4834)

20. Secondary Outcome: Mean Binocular Photopic Contrast Sensitivity With Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested binocularly (both eyes) in photopic (well-lit) conditions, with a glare source, using sine waving gratings in a computerized testing system. The photopic spatial frequencies tested were 3, 6, 12, 18 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 260 | 67
Number analyzed (log units) | 260 | 67
log units on a scale
  Spatial Frequency 3 cpd | 1.866 (0.3893) | 1.983 (0.3217)
  Spatial Frequency 6 cpd | 1.856 (0.3853) | 1.891 (0.3745)
  Spatial Frequency 12 cpd | 1.431 (0.4408) | 1.476 (0.4720)
  Spatial Frequency 18 cpd | 0.957 (0.4388) | 0.970 (0.4516)

21. Secondary Outcome: Mean Binocular Mesopic Contrast Sensitivity Without Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested binocularly (both eyes) in mesopic (low-light) conditions, without a glare source, using sine waving gratings in a computerized testing system. The mesopic spatial frequencies tested were 1.5, 3, 6, 12 cycles per degree (cpd). When a subject was unable to see the highest contrast, the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 260 | 67
Number analyzed (log units) | 260 | 67
log units on a scale
  Spatial Frequency 1.5 cpd | 1.936 (0.3442) | 1.969 (0.4236)
  Spatial Frequency 3 cpd | 2.030 (0.3306) | 2.079 (0.3129)
  Spatial Frequency 6 cpd | 1.688 (0.3922) | 1.723 (0.4132)
  Spatial Frequency 12 cpd | 0.995 (0.4098) | 0.986 (0.4300)

22. Secondary Outcome: Mean Binocular Mesopic Contrast Sensitivity With Glare
Description: Contrast sensitivity (the ability to distinguish between an object and it's background) was evaluated in a subgroup of subjects and was tested binocularly (both eyes) in mesopic (low-light) conditions, with a glare source, using sine waving gratings in a computerized testing system. The mesopic spatial frequencies tested were 1.5, 3, 6, 12 cycles per degree (cpd). When a subject was unable to see the highest contrast grating, the highest contrast score was assigned. Raw scores (0 to 9) from contrast sensitivity testing were transformed to log units. Better results are reflected by a higher numeric value.
Time Frame: 6 Months (160-210 days post second eye operative visit)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log units on a scale
Units Other Than Participants: log units
Arm/Group | IC-8™ IOL Group | Control Group
Number analyzed (Participants) | 260 | 67
Number analyzed (log units) | 260 | 67
log units on a scale
  Spatial Frequency 1.5 cpd | 1.395 (0.4280) | 1.559 (0.3979)
  Spatial Frequency 3 cpd | 1.602 (0.4527) | 1.714 (0.3955)
  Spatial Frequency 6 cpd | 1.382 (0.4254) | 1.403 (0.3575)
  Spatial Frequency 12 cpd | 0.797 (0.3951) | 0.756 (0.4223)

ADVERSE EVENTS:
Time Frame: Second eye implantation through study completion; approximately 1-year (12 months).
Description: Adverse Events (AE) were obtained through both solicited (non-directed questions) and spontaneous reports from subjects, as well as through observations by the Investigator during clinical examination. The Safety population (analysis population) includes all bilaterally implanted subjects as well as those subjects not successfully implanted with the IC-8™ IOL but for whom the IC-8™ IOL touched the eye. Ocular Adverse Events are based on a Modified Version of AAO Consensus (Masket et al., 2017).
Groups:
- Preoperative: All subjects in the safety analysis population (Intent-to-Treat population) prior to second eye implantation.
- IC-8™ IOL Group - 2nd Eye: All second eyes (study eyes) implanted with IC-8™ IOL in the IC-8™ IOL Group.
- IC-8™ IOL Group - 1st Eye: All first eyes (fellow eyes) implanted with an AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00, or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the IC-8™ IOL Group.
- IC-8™ IOL Group - Systemic: All subjects implanted with the IC-8™ IOL in the IC-8™ IOL Group.
- Control Group - 2nd Eye: All second eyes implanted with an AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00, or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the Control Group.
- Control Group - 1st Eye: All first eyes implanted with an AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00, or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the Control Group.
- Control Group - Systemic: All subjects implanted with an AcrySof® IQ SA60WF or TECNIS® aspheric monofocal ZCB00, or monofocal toric IOL (AcrySof® IQ SA6AT3, SA6AT4 or TECNIS® ZCT150 or ZCT225) in the Control Group.
Arm/Group | Preoperative | IC-8™ IOL Group - 2nd Eye | IC-8™ IOL Group - 1st Eye | IC-8™ IOL Group - Systemic | Control Group - 2nd Eye | Control Group - 1st Eye | Control Group - Systemic
All-Cause Mortality (participants affected / at risk) | 0/453 | 0/343 | 0/343 | 0/343 | 0/110 | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/453 | 6/343 | 2/343 | 22/343 | 1/110 | 1/110 | 5/110
Other Adverse Events (participants affected / at risk) | 0/453 | 264/343 | 148/343 | 114/343 | 56/110 | 55/110 | 50/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative (N=453) | IC-8™ IOL Group - 2nd Eye (N=343) | IC-8™ IOL Group - 1st Eye (N=343) | IC-8™ IOL Group - Systemic (N=343) | Control Group - 2nd Eye (N=110) | Control Group - 1st Eye (N=110) | Control Group - Systemic (N=110)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aneursysm (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart failure/Congestive heart failure (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischemic heart disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Solid tumour (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attack (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystoid Macular Edema (Eye disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular Pressure Increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iris Injury (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative (N=453) | IC-8™ IOL Group - 2nd Eye (N=343) | IC-8™ IOL Group - 1st Eye (N=343) | IC-8™ IOL Group - Systemic (N=343) | Control Group - 2nd Eye (N=110) | Control Group - 1st Eye (N=110) | Control Group - Systemic (N=110)
Abdominal pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Acute liver failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered Visual Depth Perception (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anterior Capsular Phimosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis/Atherosclerosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia/Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Bronchospasm/Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brow, Eyelid Ptosis (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Cataract Fragments in Eye Following Cataract Surgery (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract Operation Complication, Lens Dislocation (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract Subcapsular (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterization arterial normal (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ciliary Zonular Dehiscence, Vitreous Prolapse (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cold sores (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Common cold syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival Edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival Hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival abrasion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Convulsion/Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal Abrasion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Corneal Deposits, Cornea Verticillata (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal Dystrophy (Eye disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal Epithelial Defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal Epithelial Microcysts (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal stromal edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cramp(s)/Muscle spasm(s) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cystoid Macular Edema (Eye disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Damage to ligament(s) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Detached Descemet's membrane (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Detachment of retinal pigment epithelium, Retinal depigmentation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device Damage (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 32 (32) | 26 (26) | 0 (0) | 9 (9) | 9 (9) | 0 (0)
Dysphotopsia (Eye disorders) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid infection (Eye disorders) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid tumor (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Halo Vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 5 (5)
Heart failure/Congestive heart failure (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis, unspecified (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
High blood pressure/Hypertension (General disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 1 (1)
High pulmonary arterial wedge pressure (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolemia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypersensitivity/Allergic reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertension worsened (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression or protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Eye disorders) | 0 (0) | 19 (19) | 16 (16) | 0 (0) | 10 (10) | 7 (7) | 0 (0)
Iris transillumination defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 15 (15) | 7 (7) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Keratic precipitates (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low blood pressure/Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle/Tendon damage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Ocular Discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disease NOS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Polyp of nasal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior Vitreous Detachment (Eye disorders) | 0 (0) | 19 (19) | 8 (8) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 111 (111) | 48 (48) | 0 (0) | 19 (19) | 18 (18) | 0 (0)
Posterior capsule tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Punctate Keratitis (Eye disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 3 (3)
Restless legs syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal Drusen (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinal Tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swollen lymph nodes/glands (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/Thrombus (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombus (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attack (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unspecified infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Unspecified mental, emotional or behavioural problem (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Unspecified musculoskeletal problem (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Unspecified nervous system problem (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Urolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uveitis (intermediate) (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreoretinal Traction Syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Whiplash injury to neck (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the PI must provide sponsor a manuscript of such submission(s) for review, comment and approval at least 90 days prior to a planned submission for publication or presentation and that sponsor is permitted to delay any publication or presentation in specific circumstances.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03633695/Prot_SAP_000.pdf